CLINICAL TRIAL: NCT03109886
Title: Phase IIA Exploratory Study of Oral Milciclib Maleate in Patients With Unresectable or Metastatic Hepatocellular Carcinoma
Brief Title: Study of Milciclib in Patients With Unresectable/Metastatic Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDKO-125a-010; 2017-000144-18 (EudraCT Number)
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Unresectable Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma; Child-Pugh Class A
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — N,1,4,4-tetramethyl-8-((4-(4-methylpiperazin-1-yl)phenyl)amino)-4,5-dihydro-1H-pyrazolo(4,3-h)quinazoline-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Milciclib maleate (Experimental): milciclib maleate ,10, 50 and 100 mg hard gelatine capsules , 100 mg once daily, for 4 consecutive days a week in a 4-week cycle (4 days on/3 days off x q4 wks) for a total of 12 weeks (i.e. 3 cycles)
  Interventions: Drug: Milciclib maleate

INTERVENTIONS:
Drug: Milciclib maleate — 100 mg/day once daily, for 4 consecutive days a week in a 4-week cycle (4 days on/3 days off x q4 wks) for a total of 12 weeks (i.e. 3 cycles) unless patient refusal, consent withdrawal, Investigator's decision, unacceptable toxicity or death whichever occurs earlier. After the completion of three cycles, patients who, in the Investigator's judgment, are benefiting from treatment with milciclib, will resume treatment and will remain on study up to Day 180 from treatment start, unless withdrawal criteria are met earlier.
  Other Names: PHA-848125AC

SUMMARY:
The primary aim of this exploratory study is to test the safety and tolerability of milciclib when administered orally at 100 mg in patients with recurrent or metastatic Hepatocellular Carcinoma. The evaluation of the efficacy profile is a secondary objective of the study. Moreover, markers expression in tumor cells and plasma will be studied and described in association with the clinical outcome.

Eligible patients will receive milciclib orally on a daily schedule for 4 consecutive days a week in a 4-week cycle (4 days on/3 days off x q4 wks) for a total of 12 weeks (i.e. 3 cycles) unless patient refusal, consent withdrawal, Investigator's decision, unacceptable toxicity or death whichever occurs earlier.

At the end of Cycle 3, treatment will be stopped, and based on the results of the tumor assessment performed on Day 90 (±3 days) from treatment start, patients will be followed as here below detailed:

* patients with Complete Response (CR)/Partial Response (PR)/Stable Disease (SD) will be followed for safety until 30 days from last dose intake (or until a new anticancer therapy starts, whichever occurs earlier) and will be assessed for efficacy in the follow-up period up to Day 180 from treatment start;
* patients with progressive disease will be followed only for safety until 30 days from last dose intake (or until a new anticancer therapy starts, whichever occurs earlier).

After the completion of three cycles, patients who, in the Investigator's judgment, are benefiting from treatment with milciclib, will resume treatment and will remain on study up to Day 180 from treatment start, unless withdrawal criteria are met earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of HCC, confirmed by histology or radiology according to American Association for the Study of Liver Diseases/European Association for the Study of the Liver (AASLD/EASL) criteria prior to the start of the investigational product. Imaging characteristics should be retrieved from at least a 3-phase liver protocol CT or MRI with target tumor lesion(s) demonstrating arterial hyper-enhancement and wash-out in the venous phase;
* Tumor stages eligible for the study are defined as:

  1. HCC within the Barcelona Clinic Liver Cancer (BCLC) stage C. In case of portal vein thrombosis (PVT) an associated target lesion in the liver parenchyma should be clearly defined. PVT without associated target lesion are not eligible to the study;
  2. Untreatable post-chemoembolization (TACE) or post-radioembolization (TARE) progression defined as BCLC stage B or C with radiographic progression according to mRECIST after TACE or TARE not eligible for further surgical or loco-regional therapy;
  3. Recurring HCC non eligible for pre-transplant downstaging protocols or for resection;
* Patients must have failed sorafenib treatment or be intolerant to sorafenib or actively refusing sorafenib

  1. Failing sorafenib treatment is defined if after ≥ 14 days of therapy (not necessarily consecutive) radiology progression is ascertained according to mRECIST;
  2. Intolerant to sorafenib treatment is defined as a sorafenib related Grade 2 or greater adverse event (CTC-AE) that continues or recurs after sorafenib treatment interruption for 7 days or dose reduction;
  3. Active refusal should be documented by a written and signed patient declaration to be filed in the clinical records;
* Child-Pugh score ≤ 6 (class A);
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Local or loco-regional therapy (i.e., surgery, radiation therapy, hepatic arterial embolization, chemoembolization, radioembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) must have been completed ≥4 weeks prior to study entry with documentation of progressive or recurrent disease;
* Signed and dated Investigational Review Board/Independent Ethics Committee (IRB/IEC) approved Informed Consent/Genetic Consent.

Exclusion Criteria:

* Prior use of any systemic anti-cancer therapy (including experimental agents and immunotherapy) except for sorafenib and second line treatment with regorafenib discontinued for intolerance within 14 days;
* Known fibrolamellar HCC or mixed hepato-cholangiocarcinoma;
* Grade 3 oesophageal varices, regardless of previous bleeding episodes on endoscopy performed no more than in the last 12 months;
* Clinical meaningful ascites defined as CTCAE Grade≥2. Patient who have been on a stable medication regimen for at least 2 months to manage ascites are eligible if they show no ascites at the clinical examination. Patients with clinically undetectable ascites who are Child A with detectable ascites at CT/MRI are eligible to the protocol;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Overall Safety Profile | From Informed Consent signature to 30 days after last dose intake up to Day 180 from treatment start
  Overall safety profile, evaluated on the basis of laboratory (i.e. hematology and blood chemistry, urinalysis, vital signs, ophthalmologic examinations) and adverse events emerging during the trial, will be determined. The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 will be used for the severity grading of adverse events and of hematological and blood chemistry abnormalities

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At screening; During treatment at Day 45 and 90; During follow up at Day 180 for patients not progressed at previous assessments
  Confirmed CR. The objective tumor assessment will be made according to the modified Response Evaluation Criteria In Solid Tumors (mRECIST) criteria for Hepatocellular Carcinoma (HCC). Conventional RECIST 1.1 will be also assessed. ORR will be assessed locally and confirmed by an Independent Central Review.
Objective Response Rate (ORR) | At screening; During treatment at Day 45 and 90; During follow up at Day 180 for patients not progressed at previous assessments
  Confirmed PR. The objective tumor assessment will be made according to the modified Response Evaluation Criteria In Solid Tumors (mRECIST) criteria for Hepatocellular Carcinoma (HCC). Conventional RECIST 1.1 will be also assessed. ORR will be assessed locally and confirmed by an Independent Central Review.
Progression-Free Survival (PFS) | From treatment start to date of progression assessed on Day 45, 90 or 180 or to date of death if before day 180
  PFS is evaluated since study treatment start to progression, based on mRECIST tumor assessment, or death for any causes.
Time to Progression (TPP) | From treatment start to date of progression assessed on Day 45, 90 or 180 or to date of death if before day 180
  TPP is evaluated since study treatment start to progression, based on mRECIST tumor assessment or death due to disease progression in the absence of previous documented Progression Disease (PD).
TPP-3 months | Based on tumor assessment at or after 3 months from treatment start
  Proportion of evaluable patients known to be alive and progression free based on mRECIST tumor assessment at ≥ 3 months since study treatment start out of the total number of evaluable patients (TTP-3 months)
Duration of overall Response (DoR) | Based on assessments performed on Day 45, 90 or 180 or date of death if before day 180
  DoR is measured from the time measurement criteria are first met for CR/PR based on mRECIST tumor assessment, until the first date that recurrence or PD is objectively documented or death date due to tumor progression in the absence of previous documented PD.

CONTACTS AND LOCATIONS:
Overall Officials: Fayez M Hamzeh, MD, Study Chair — Tiziana Life Sciences LTD; Angelo Sangiovanni, MD, PHD, Principal Investigator — Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico - Milano, Italy; Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas - Rozzano (MI), Italy
Locations (14):
- Greece (4):
  - Ippokrateio General Hospital of Athens, Athens
  - Laiko General Hospital of Athens, Athens
  - General University Hospital of Larissa, Larissa
  - University General Hospital of Thessaloniki - AHEPA, Thessaloniki
- Israel (4):
  - Rambam Health Corporation, Haifa
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - The Sheba Academic Medical Center Hospital - Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Istituto Clinico Humanitas, Rozzano, MI
  - AOU S. Orsola Malpighi Bologna, Bologna
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Policlinico di Modena, Modena
  - A.O.U. Federico II, Napoli
  - A.O. U. Policlinico Paolo Giaccone, Palermo

IPD SHARING:
Plan to Share IPD: No